CLINICAL TRIAL: NCT04681443
Title: Factors Affecting Outcomes of Crystallized Phenol Application in the Treatment of Pilonidal Sinus Disease
Brief Title: Crystallized Phenol Treatment in Pilonidal Sinus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gulhane Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Suleyman Utku Celik, Principal Investigator, Gulhane Training and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Gulhane2020-146
Record Dates: First submitted 2020-12-17; First posted 2020-12-23 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Pilonidal Sinus of Natal Cleft; Pilonidal Sinus Without Abscess
Keywords: pilonidal disease; crystallized phenol; outcomes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Successful treatment (Active Comparator): Patients with successfully treated pilonidal sinus disease
  Interventions: Drug: Crystallized phenol application
- Treatment failure (Active Comparator): Pilonidal sinus disease patients with treatment failure
  Interventions: Drug: Crystallized phenol application

INTERVENTIONS:
Drug: Crystallized phenol application — Crystallized phenol application into the sinus tract

SUMMARY:
Pilonidal sinus disease is an acquired disorder of the natal cleft and its incidence is reported as 6 in 100,000. Although there are many opinions regarding the treatment of pilonidal sinus disease in the literature, surgery is the main treatment method. Regardless of the treatment protocol, this disease has a certain risk of recurrence. Therefore, the ideal treatment procedure for the pilonidal disease should be simple to perform, should allow patients to return earlier to work, should be associated with minimal pain, and should minimize financial cost.

Phenol application into the pilonidal sinus is an additional nonoperative adjunct to treatment. This method is typically used after all hair and debris have been removed or curetted from the sinus, and it helps to eliminate granulation tissue and further debris formation. The injection is followed by hair control and strict hygiene. The use of phenol causes an intense inflammatory reaction which destroys the epithelial lining, and care should be taken to protect the surrounding skin. Pain is intense and may require inpatient admission for pain control but success rates have been reported to range from 60% to 95%. However, it is difficult to know which patients can expect enough benefit from phenol application.

The aim of the study is to evaluate the factors affecting the outcomes of patients with the pilonidal disease treated with crystallized phenol and to evaluate long-term recurrence rates of pilonidal disease treated with crystallized phenol.

DETAILED DESCRIPTION:
Pilonidal sinus disease is an acquired disorder of the natal cleft and its incidence is reported as 6 in 100,000. Although there are many opinions regarding the treatment of pilonidal sinus disease in the literature, surgery is the main treatment method. Regardless of the treatment protocol, this disease has a certain risk of recurrence. Therefore, the ideal treatment procedure for the pilonidal disease should be simple to perform, should allow patients to return earlier to work, should be associated with minimal pain, and should minimize financial cost.

Phenol application into the pilonidal sinus is an additional nonoperative adjunct to treatment. This method is typically used after all hair and debris have been removed or curetted from the sinus, and it helps to eliminate granulation tissue and further debris formation. The injection is followed by hair control and strict hygiene. The use of phenol causes an intense inflammatory reaction which destroys the epithelial lining, and care should be taken to protect the surrounding skin. Pain is intense and may require inpatient admission for pain control but success rates have been reported to range from 60% to 95%. However, it is difficult to know which patients can expect enough benefit from phenol application.

In this study, the procedure will be performed on an outpatient basis and the treatment procedure will be performed in the prone position. Previously shaved sacrococcygeal area will be cleaned with an antiseptic solution and local anesthesia will be achieved using 2% lidocaine (1:100,000 adrenaline). After sinuses are dilated with a mosquito clamp; hair, debris, and granulation tissue will be removed from the sinus tracts using a curved surgical forceps and the tracts will be curetted using a straight curette. Following the protection of the skin surrounding the sinus openings with a pomade and the perianal area with a sponge, the sinus cavity will be sclerosed using crystallized phenol. Crystallized phenol will be inserted into the sinus tract from the dilated sinus opening with a clamp until the tract is full. This procedure will repeat twice and each phenol particles will remain in sinus about one minute, and then will be removed by applying pressure. Consequently, the procedure will be completed after dressing and the patient will be sent home by prescribing an analgesic pill (paracetamol 500 mg) to use only when required.

After the patients are divided into two groups: (1) those successfully treated and (2) those with treatment failure, descriptive statistics will be presented as the means +/- standard deviations (SDs), medians and interquartile ranges (IQRs), and frequencies (%). Examinations of normal distribution assumptions for continuous variables will be visually assessed with quartile-quartile plots and histograms and confirmed with the Shapiro-Wilk test. Associations between variables will be evaluated using the Mann-Whitney U and Student's t tests (for continuous variables) or Pearson's chi-square and Fisher exact tests (for categorical variables), where appropriate.

The association of treatment success with demographics, symptom duration, and pilonidal sinus features such as the number and location of the sinuses, the amount of hair inside the sinus, the volume of the sinus tract, and the length of sinus tract will be analyzed with logistic regression analysis. First, each covariate will be analyzed in a univariate model, and all variables with p-value less than 0.20 will be included in the final multivariate logistic regression model to determine independent factors. Odds ratios (ORs) of statistically significant predictors will be presented with 95% confidence intervals (CIs). P values lower than 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptoms due to chronic primary or recurring pilonidal sinus disease interfering with daily life
* Patients giving written informed consent
* Patients who can be contacted by e-mail or telephone
* Patients aged 18 years and older

Exclusion Criteria:

* Patients with no or minimal symptoms related to pilonidal sinus disease
* Patients with an acute pilonidal abscess or complex, multiple recurrent pilonidal diseases
* Patients who could not be contacted during the follow-up period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Short-term recurrence rate | 30 days
  To evaluate short-term recurrence rates of pilonidal disease treated with crystallized phenol.
Healing time | 1 year
  To evaluate the mean time from initial treatment to healing the sinus

SECONDARY OUTCOMES:
Long-term recurrence rates | 1 year
  To evaluate long-term recurrence rates of pilonidal disease treated with crystallized phenol.

CONTACTS AND LOCATIONS:
Overall Officials: Suleyman Utku Celik, MD, Principal Investigator — Gulhane Training and Research Hospital
Locations (1):
- Gulhane Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Kayaalp C, Olmez A, Aydin C, et al. Investigation of a one-time phenol application for pilonidal disease. Med Princ Pract 2010;19(3):212-5. — https://pubmed.ncbi.nlm.nih.gov/20357505/
- See also: Dag A, Colak T, Turkmenoglu O, et al. Phenol procedure for pilonidal sinus disease and risk factors for treatment failure. Surgery 2012; 151(1):113-7. — https://pubmed.ncbi.nlm.nih.gov/21982072/
- See also: Steele SR, Perry WB, Mills S, et al. Practice parameters for the management of pilonidal disease. Dis Colon Rectum 2013; 56(9):1021-7.. doi: 10.1097/DCR.0b013e31829d2 — https://pubmed.ncbi.nlm.nih.gov/23929010/